CLINICAL TRIAL: NCT01632397
Title: Optimizing Antiretroviral-Based Prevention by Enhancing PrEP Adherence in MSM
Brief Title: Pre-exposure Prophylaxis Adherence Intervention for MSM
Acronym: PrEPare
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fenway Community Health (Other)
Responsible Party: Principal Investigator, Kenneth H. Mayer, MD, Medical Research Director, Co-Chair of The Fenway Institute, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34MH095584-01 (NIH)
Record Dates: First submitted 2012-05-08; First posted 2012-07-02 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Medication Adherence
Keywords: PrEP; HIV; Adherence; MSM; Men having sex with men
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-based counseling (Experimental): Cognitive behavioral based intervention to promote PrEP adherence.
  Interventions: Behavioral: CBT-based counseling
- Health education and supportive counseling (Active Comparator): Time matched supportive counseling
  Interventions: Behavioral: Health education and supportive counseling

INTERVENTIONS:
Behavioral: CBT-based counseling — Cognitive Behavior Therapy for PrEP adherence
  Arms: CBT-based counseling
Behavioral: Health education and supportive counseling — Time matched general supportive therapy of the type commonly available from community therapists.
  Arms: Health education and supportive counseling

SUMMARY:
Following formative work, the proposed study is an open-label, pilot, randomized, two arm trial where subjects will receive pre-exposure prophylaxis (PrEP) for 6 months and either a cognitive-behavioral based adherence intervention or health education with supportive counseling.

ELIGIBILITY:
Inclusion Criteria:

* male sex at birth
* being 18 years old or older
* testing HIV-negative at screening
* evidence of high risk for HIV acquisition defined by having unprotected anal sex (insertive or receptive) with an HIV-positive male partner OR at least a total of three episodes of unprotected anal sex with at least two partners in the last three months
* medically cleared to take the study drug (ambulatory performance >=60 on Karnofsky scale, adequate renal function, negative glucose and protein in urine, adequate hepatic function, adequate hematologic function)
* able to understand and speak English (for consenting and counseling).

Exclusion Criteria:

* participants who are not able to consent due to psychiatric or cognitive concerns
* those who have already been prescribed PrEP
* having a history of or current medical conditions that would preclude taking the study drug (e.g., previously diagnosed active and serious infections, acute or chronic hepatitis B, history of pathological bone fractures not related to trauma)
* receiving ongoing therapy with ART, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion, or other investigational agents
* receiving or possibly receiving antiretroviral drugs for an anti-HIV vaccine in a clinical trial
* active alcohol or drug use that would interfere with study participation
* having other conditions (based on opinion of investigator or designee) that would preclude informed consent, make the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Adherence to PrEP over time | At each of the 7 study visits post PrEP perscrition spread over the duration of the study (up to six months)
  This is primarily a feasiblity pilot RCT. However, the primary eventual endpoint is PrEP adherence measured daily via electronic medication adherence monitoring (Wisepill™).

SECONDARY OUTCOMES:
Sexual Risk Compensation | At each of the 9 study visits spread over up to six months.
  This is primarily a feasiblity RCT. Sexual risk compensation is defined as a potential change in sexual risk taking behaviors (unprotected anal sex). This is measured daily with text message assessments for sexual risk as well as at each study visit with self-report measure(s).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mayer, MD, Principal Investigator — Fenway Health
Locations (1):
- The Fenway Institute, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21091279